CLINICAL TRIAL: NCT01828801
Title: Cross-Sectional, Multi-Center Evaluation of 8 Year Metal Ion Trends for Pinnacle MoM System Used in Primary Hip Arthroplasty
Brief Title: Pinnacle Metal-on-Metal 522 Post-Market Surveillance Study
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 10017
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-05

CONDITIONS: Pinnacle Metal-on-Metal; Revised Pinnacle Metal-on-Metal; Adverse Local Tissue Reaction; Metal Ions; Total Hip Arthroplasty
Keywords: Adverse Local Tissue Reaction; Metal Ions; Serum; Whole Blood; Metal-on-Metal; Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and serum samples are retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Pre-Op: Pre-operative patients who will undergo a total hip replacement.
- 1 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 1 year post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 2 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 2 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 3 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 3 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 4 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 4 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 5 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 5 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 6 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 6 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 7 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 7 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal
- 8 year post-op: Patients that underwent a Pinnacle Metal-on-Metal (MoM) total hip replacement (THR) and at the time of enrollment, based on their date of surgery, were 8 years post-operative . Alternatively these are patients who have had their Pinnacle Metal-on-Metal hip revised but if they were not revised, would have fallen into this time point.
  Interventions: Device: Pinnacle Metal-on Metal

INTERVENTIONS:
Device: Pinnacle Metal-on Metal — All patients that are post-operative will have undergone total hip arthroplasty with the Pinnacle Metal-on-Metal device
  Other Names: Pinnacle MoM; Ultamet
  Groups: 1 year post-op; 2 year post-op; 3 year post-op; 4 year post-op; 5 year post-op; 6 year post-op; 7 year post-op; 8 year post-op

SUMMARY:
The purpose of this clinical study is to evaluate blood metal ion levels as a function of time of implantation for the Pinnacle Acetabular MoM system.

ELIGIBILITY:
Inclusion Criteria:

1. Able to (or capable of) provide written, voluntary consent to participate in the clinical investigation
2. Is willing and able to return for all protocol defined clinic visits
3. Subject has a combination of the following implants in the study hip (unless in pre-op cohort):

   1. Pinnacle acetabular shell with or without Gription TM porous coating
   2. M-specification cobalt-chrome femoral head or aSphere M-specification cobalt-chrome femoral head
   3. Ultamet metal insert
   4. One of the following stems

   i. S-ROM ii. Corail iii. Tri-Lock iv. AML v. Summit vi. Prodigy vii. C-Stem
4. Subject has high quality films available for review that were taken within 12 months of the primary surgery of the following views:

   1. Standing AP-Pelvis
   2. Standing AP-Proximal Femur (if this view is not available but the AP-Pelvis shows the entire implant and greater trochanter, that is also acceptable)
   3. Lauenstein Lateral Proximal Femur (Lateral-Femur)

Exclusion Criteria:

1. The subject refuses to allow their medical records to be inspected by the Sponsor, representatives of the Sponsor, the medical office staff and/or representatives from FDA
2. The implanted hip components in the study hip (exclusive of cement), are not all DePuy components (unless in pre-op cohort)
3. The primary procedure occurred greater than 8 (eight) years ago (unless in pre-op cohort)
4. FOR PRE-OPERATIVE COHORT ONLY: the subject has a MoM contralateral hip
5. FOR PRE-OPERATIVE COHORT ONLY: the subject is undergoing a revision of the Ipsilateral hip

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have undergone a total hip arthroplasty with the Pinnacle Metal-on-Metal device within the past 8 years.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Chromium serum ion level across time intervals | Pre-operatively through 8 years
  To compare the chromium serum ion levels in the patient population from pre-operatively through 8 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (pre-operatively through 8 years post-operatively) will be a different cohort of patients.
Change in Chromium whole blood ion level across time intervals | Pre-operatively through 8 years
  To compare the chromium whole blood ion levels in the patient population from pre-operatively through 8 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (pre-operatively through 8 years post-operatively) will be a different cohort of patients.
Change in Cobalt serum ion level across time intervals | Pre-operatively through 8 years
  To compare the cobalt serum ion levels in the patient population from pre-operatively through 8 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (pre-operatively through 8 years post-operatively) will be a different cohort of patients.
Change in Cobalt whole blood ion level across time intervals | Pre-operatively through 8 years
  To compare the cobalt whole blood ion levels in the patient population from pre-operatively through 8 years post-operatively in a 1-way ANOVA. This is a cross-sectional study so each time interval (pre-operatively through 8 years post-operatively) will be a different cohort of patients.

SECONDARY OUTCOMES:
Poolability of data across stem types | Pre-operatively through 8 years post-operatively
  Within each of the primary analyses, the poolability of data across stem types will be confirmed with a 2-way ANOVA model in which both time interval and stem type are independent variables.
Incidence of adverse local tissue reaction (ALTR) | Pre-operatively through 8 years post-operatively
  To determine trends in the incidence of ALTR over time.
Implant survivorship | Through 8 years post-operatively
  To determine implant survivorship, where an implant is considered to be surviving when none of the total hip replacement (THR) system components have been removed or replaced, so that the original system with metal-on-metal (MoM) articulating surfaces remains intact. Implant survivorship will be analyzed in two ways: 1) for all revisions (for any reason) and 2) for revisions due to ALTR.
To identify the incidence of ALTR among unrevised subjects | Through 8 years post-operatively
  To identify the incidence of ALTR among unrevised subjects through physical examination and imaging.
Ion levels among revised subjects | Pre-operatively through 8 years post-operatively
  To compare cobalt and chromium ion level (prior to revision) vs. baseline for subjects who are revised.
Harris Hip and HOOS analysis for pain, function and total score | Though 8 years post-operatively
  To identify the incidence of pain or functional symptoms among unrevised subjects with a Harris Hip and HOOS evaluation. To compare cobalt and chromium ion levels for unrevised subject who are exhibiting pain or functional symptoms vs. unrevised subjects who are not exhibiting pain or functional symptoms.
To determine the association of adverse events with elevated ion levels | Through 8 years post-operatively
  To investigate the association of adverse events with elevated cobalt and chromium ion levels. For each respective adverse event, to compare cobalt and chromium ion levels for subjects who have vs. subjects who have not exhibited the adverse event. For each respective adverse event category, to present summary statistics of cobalt and chromium ion levels for subjects who have vs. subjects who have not exhibited the adverse event, stratified by post-op time cohort.
Trending | Through 8 years post-operatively
  Trends (over time since initial implant) will be evaluated for: 1) revisions (survivorship), 2) adverse events, 3) pain or functional symptoms (via Harris Hip and HOOS evaluations), 4) incidence of ALTR in unrevised subjects
Patient history and demographics and association with outcomes | Throughout 8 years post-operatively
  Patient demographic and subject history will be evaluated for association with: 1) higher metal ion levels and 2) risk of revision.
Modes and causes of implant failure | Through 8 years post-operatively
  To evaluate modes and causes of implant failure based on an analysis of reasonably available explanted retrieved devices.
Metal ion levels and association with reason for revision | Through 8 years post-operatively
  To compare cobalt and chromium levels across the different reasons for revision.
Comparison of metal ion levels across subjects with vs. without ALTR | Through 8 years post-operatively
  Cobalt and Chromium ion levels will be compared for unrevised subjects who were not diagnosed with an ALTR vs. unrevised subject who were diagnosed with an ALTR.
Ion level vs. baseline for ALTR subjects | Through 8 years post-operatively
  To compare cobalt and chromium ion level vs. baseline for subject who are diagnosed with ALTR.
Ion level change from first measurement for ALTR subjects | Through 8 years post-operatively
  Cobalt and chromium ion levels will be compared from first measurement to the time of revision (prior to revision) or the time of last follow-up visit in the study, whichever comes first, for subjects who are diagnosed with an ALTR.

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Panozzo, BS, Study Director — DePuy Synthes Joint Reconstruction
Locations (8):
- United States (8):
  - Orange, California
  - Fort Collins, Colorado
  - Lone Tree, Colorado
  - Syracuse, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnatti, Ohio
  - Austin, Texas